CLINICAL TRIAL: NCT05180669
Title: Reward-based Technology to Improve Opioid Use Disorder Treatment Initiation After an ED Visit - Phase 2
Brief Title: Reward-based Technology to Improve OUD Treatment
Acronym: OARSCM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was impacted by a massive epidemiological shift that led to reduced rates of presentation to the ED for opioid overdose. Despite more than a year of adjusting protocols and site expansion, we were not able to meet study enrollment goals.
Sponsor: Q2i, LLC (Industry)
Collaborators: University of Massachusetts, Worcester (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H00017879-2; R42DA049448 (NIH)
Record Dates: First submitted 2021-10-20; First posted 2022-01-06 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder
Keywords: Substance Use Disorder; Opioid Use Disorder; Contingency Management; Medication for opioid use disorder; Medication-assisted treatment
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Both groups will be enrolled at the same time through, with group designated by randomization, and monitored through the 12-week RCT as well as follow ups at 1-, 3-, and 6-months post enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OARSCM (Experimental): OARSCM (n = 21) patients will receive the same TAU procedures described above. They will also earn chances for prizes, with the same targeted behaviors, escalation of chances for prizes for each targeted behavior in a row, and reset criteria described. Briefly, for scheduling a MOUD treatment intake, patients will earn 2 chances for prizes. Chances for prizes will increase by 2 chances with documentation of each targeted behavior in a row up to a maximum of 10 draws/targeted behavior. With 38 targeted behaviors (schedule MOUD intake, complete intake, 12 opioid-negative urine toxicology/week over 12 weeks plus bonuses for cocaine-negative tests, and 12 group/individual therapy/week over 12 weeks), patients can earn up to 252 chances for prizes during the 12-week RCT.
  Interventions: Other: OARSCM Software Application
- TAU with MyMAT (Sham Comparator): TAU (n = 20) In the acute care setting, the Behavioral Health Service provides SBIRT for substance use disorders, including OUD. They provide SBIRT as part of TAU, including a warm handoff to an outpatient MOUD treatment with a scheduled outpatient appointment, optimally within 48 hours of the ED visit. TAU outpatient suboxone treatment consists of urine toxicology screening, group/individual therapy, and MOUD prescription continent on drug-negative urine toxicology. Treatment visits are typically weekly in weeks 1-4 and then taper over time, to every other week in weeks 5-8, and monthly in weeks 9-12 and after. Nonadherence can lead to increased frequency/intensity of therapy and urine toxicology until the patient stabilizes. If increased frequency/intensity is unsuccessful, patients may be referred to detoxification and subsequently re-admitted to outpatient care when appropriate. Patients will receive MyMAT a mobile application with educational content regarding MOUD treatment.
  Interventions: Other: MyMAT Software Application

INTERVENTIONS:
Other: OARSCM Software Application — Access is granted to participants for 12 weeks to the OARSCM platform which includes reinforcements for meeting MOUD treatment goals.
  Other Names: Opioid Addiction Recovery Support - Contingency Management (OARSCM)
  Arms: OARSCM
Other: MyMAT Software Application — Access is granted to the MyMAT mobile application for 12 weeks which provides educational content regarding MOUD treatment.
  Other Names: MyMAT
  Arms: TAU with MyMAT

SUMMARY:
Millions of people in the US misuse opioids each year. Medication assisted treatment (MAT) for opioid use disorder (OUD) is highly efficacious, but only a fraction of OUD persons access MAT, and treatment non-adherence is common and associated with poor outcomes. This project will utilize a digital mobile platform, Opioid Addiction Recovery Support with contingency management (OARSCM), to increase MAT treatment initiation and adherence among OUD patients recruited from emergency departments and inpatient acute care.

DETAILED DESCRIPTION:
Millions of people in the US misuse opioids each year, leading to thousands of deaths and costing billions of dollars in total economic burden. Medication assisted treatment (MAT) for opioid use disorder (OUD) is highly efficacious, but only a fraction of OUD persons access MAT, and treatment non-adherence is common and associated with poor outcomes. This STTR Fast Track proposal is designed to increase rates of Suboxone (buprenorphine/naloxone) treatment initiation and adherence among OUD patients recruited from emergency and inpatient acute care. To accomplish these aims, the project will enhance the Opioid Addiction Recovery Support (OARS), an existing Q2i company technology, with a new evidence-based reward, contingency management (CM) function. CM interventions systematically reward (reinforce) specific behaviors like treatment initiation and adherence with therapy attendance and drug-free urine tests and are highly efficacious. An OARS solution enhanced with a CM component (OARSCM) that allows for the automatic calculation, delivery, and redemption of rewards contingent on objective evidence of treatment behaviors may be key to improving Suboxone initiation and adherence. In Phase 1 of this proposal, the existing OARS clinician portal and patient mobile application will be modified to accommodate entry into the software system from an acute care setting and to automatically manage and deliver rewards to create OARSCM using patient-centered design principles. Focus groups with OUD patients and other key stakeholders will inform design. Primary usability outcomes will be examined, and the program iteratively updated. After meeting milestones, there was a proof-of-concept pilot of usability, acceptability, and effects on initial behavior targets with approximately 20 patients and at least 4 providers. After meeting milestones, this RCT will follow, in which acute care OUD patients appropriate for outpatient Suboxone (N = 102) are recruited and allocated to one of two study conditions: 1) treatment as usual (TAU) with MyMAT, comprised of screening, brief intervention, referral to treatment by a trained clinician, and an educational mobile app (MyMAT), 2) OARSCM. The active intervention window for the two intervention groups will be 12 weeks. Patients will be onboarded prior to discharge from acute care. In the outpatient Suboxone setting, data on treatment adherence and opioid use will be captured from clinical records for six months. Telephone follow-up assessments and vital statics registry reviews will be at month 1, month 3 (end-of-study intervention period), and month 6. Primary Suboxone treatment initiation outcomes will be completing the Suboxone intake. Primary Suboxone treatment outcomes will be sustained abstinence at Month 6 and longest duration of abstinence. Analysis will examine data on cost avoidance and cost savings through reduced acute care visits between study conditions.

ELIGIBILITY:
Inclusion Criteria:

1. >= 18 years old
2. Presenting for acute care at UMass University and Memorial hospitals, including EDs, inpatient medical units, or inpatient behavioral health units for opioid addiction related health complaints, including opioid overdose, opioid related medical consequences, opioid intoxication or withdrawal syndromes, and/or seeking help for OUD
3. Presence of a current DSM-V opioid use disorder (OUD), mild to severe
4. Medically appropriate for outpatient Suboxone treatment, as judged by the treating clinician and behavioral health consultant or toxicologist working with the patient clinically

Exclusion Criteria:

1. Persistent altered mental status (not alert, not oriented, psychotic).
2. Not interested or willing to participate in Suboxone treatment
3. Best referral site is NOT one of the study's partner clinics in the central MA region, which will be outpatient MAT clinics and primary care within the UMass system and the three other primary facilities outside of the UMass system.
4. Unwilling to use the OARSCM app (if assigned)
5. Does not have access to their own smartphone with at least iOS 7.1 or Android 4.2, the minimal technology required to run the app, or not willing to access clinic-dedicated computer to access the program
6. Currently in state custody or pending legal action that might lead to imprisonment
7. Cannot paraphrase the study requirements
8. Does not read or speak English
9. Does not reside in the central MA region
10. Already enrolled into the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Davis-Martin, PhD, Study Director — University of Massachusetts Chan Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all individual participant data (IPD) that underlie published results.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available starting 6 months after publication of results.
Access Criteria: Deidentified data will be accessible to researchers who wish to conduct analyses not reported in prior publications. The study principal investigator will review any request for data to ensure no overlapping analyses. Deidentified data will be shared via secure, HIPAA-compliant data transfers.

REFERENCES:
- See also: Webpage for OARSCM solution — https://q2i.com/oars-cm/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals with OUD presenting to an acute care setting were approached to participate in the study between August 2022 and September 2024. Those who met the eligibility criteria and confirmed their interest in participating in the study were enrolled. The first participant was enrolled November 18, 2022 and the last patient was enrolled July 9, 2024.
Pre-assignment Details: Of the 3,006 individuals with OUD who were approached, 84 were eligible and 41 agreed to participate in the study. These 41 participants were then randomized to OARSCM (21 participants) or TAU MyMAT (20 participants).
Period: Overall Study
Arm/Group | OARSCM | TAU With MyMAT
Started | 21 | 20
1-month Follow-up | 2 | 0
3-month Follow-up | 1 | 0
6-month Follow-up | 0 | 0
Completed | 0 | 0
Not Completed | 21 | 20
Not completed — Lost to Follow-up | 21 | 20

BASELINE CHARACTERISTICS:
Groups:
- OARSCM: OARSCM (n = 51) patients will receive the same TAU procedures described above. They will also earn chances for prizes, with the same targeted behaviors, escalation of chances for prizes for each targeted behavior in a row, and reset criteria described. Briefly, for scheduling a MOUD treatment intake, patients will earn 2 chances for prizes. Chances for prizes will increase by 2 chances with documentation of each targeted behavior in a row up to a maximum of 10 draws/targeted behavior. With 38 targeted behaviors (schedule MOUD intake, complete intake, 12 opioid-negative urine toxicology/week over 12 weeks plus bonuses for cocaine-negative tests, and 12 group/individual therapy/week over 12 weeks), patients can earn up to 252 chances for prizes during the 12-week RCT.
  OARSCM Software Application: Access is granted to participants for 12 weeks to the OARSCM platform which includes reinforcements for meeting MOUD treatment goals.
- TAU With MyMAT: TAU (n = 51) In the acute care setting, the Behavioral Health Service provides SBIRT for substance use disorders, including OUD. They provide SBIRT as part of TAU, including a warm handoff to an outpatient MOUD treatment with a scheduled outpatient appointment, optimally within 48 hours of the ED visit. TAU outpatient suboxone treatment consists of urine toxicology screening, group/individual therapy, and MOUD prescription continent on drug-negative urine toxicology. Treatment visits are typically weekly in weeks 1-4 and then taper over time, to every other week in weeks 5-8, and monthly in weeks 9-12 and after. Nonadherence can lead to increased frequency/intensity of therapy and urine toxicology until the patient stabilizes. If increased frequency/intensity is unsuccessful, patients may be referred to detoxification and subsequently re-admitted to outpatient care when appropriate. Patients will receive MyMAT a mobile application with educational content regarding MOUD treatment.
  MyMAT Software Application: Access is granted to the MyMAT mobile application for 12 weeks which provides educational content regarding MOUD treatment.
- Total: Total of all reporting groups
Arm/Group | OARSCM | TAU With MyMAT | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 40
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 15 | 12 | 27
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Outpatient Intake Scheduled - Phase 2 RCT
Description: Percentage of patients who schedule an outpatient Suboxone intake prior to discharge from acute care
Time Frame: 1 timepoint - Before patients are discharged from acute care at the time of study enrollment
Population: All enrolled participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | OARSCM | TAU With MyMAT
Number analyzed (Participants) | 21 | 20
Participants
  Yes | 12 | 8
  No | 9 | 12
Statistical Analysis 1: Comparison: OARSCM vs TAU With MyMAT; Test type: Superiority; p = 0.272, Chi-squared — Statistical significance was set at p<0.05

2. Primary Outcome: Percent Outpatient Intakes Completed - Phase 2 RCT
Description: Percentage of patients who complete their outpatient Suboxone intake
Time Frame: Typically, within ~48 hours of discharge from acute care
Population: All enrolled participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | OARSCM | TAU With MyMAT
Number analyzed (Participants) | 21 | 20
Participants
  Yes | 5 | 4
  No | 16 | 16
Statistical Analysis 1: Comparison: OARSCM vs TAU With MyMAT; Test type: Superiority; p = 0.768, Chi-squared — Statistical significance was set at p<0.05

3. Secondary Outcome: Sustained Abstinence - Phase 2 RCT (Month 1)
Description: Proportion of participants with sustained abstinence (composite of biochemical & self-report data) from opioids
Time Frame: 1 month from participant's enrollment
Population: Participants who did not answer the follow-up call were considered lost to follow-up and assigned the worse possible outcome (i.e., yes, participant used opioids in past 30 days). Two OARSCM participants, one of which terminated the interview before completion, and zero TAU with MyMAT participants did the 1-month follow-up interview.
Measure: Count of Participants; unit: Participants
Arm/Group | OARSCM | TAU With MyMAT
Number analyzed (Participants) | 2 | 0
Participants
  Yes | 2 | 0
  No | 0 | 0

4. Secondary Outcome: Sustained Abstinence - Phase 2 RCT (Month 3)
Description: Proportion of participants with sustained abstinence (composite of biochemical & self-report data) from opioids
Time Frame: 3 months from participant's enrollment
Population: Participants who did not answer the follow-up call were considered lost follow-up and assigned the worse possible outcome (i.e., yes, participant used opioids in past 30 days). One OARSCM participant and zero TAU with MyMAT participants did the 3-month follow-up interview.
Measure: Count of Participants; unit: Participants
Arm/Group | OARSCM | TAU With MyMAT
Number analyzed (Participants) | 1 | 0
Participants
  Yes | 1 | 0
  No | 0 | 0

5. Secondary Outcome: Sustained Abstinence - Phase 2 RCT (Month 6)
Description: Proportion of participants with sustained abstinence (composite of biochemical & self-report data) from opioids
Time Frame: 6 months from participant's enrollment
Population: Participants who did not answer the follow-up call were considered lost follow-up and assigned the worse possible outcome (i.e., yes, participant used opioids in past 30 days). Zero participants from both arms did the 6-month follow-up interview.
Arm/Group | OARSCM | TAU With MyMAT
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Longest Duration of Abstinence - Phase 2 RCT (Month 1)
Description: Longest duration of consecutive days of abstinence (composite of biochemical & self-report data)
Time Frame: 1 month from participant's enrollment
Population: Participants who did not answer the follow-up call were considered lost to follow-up and assigned the worse possible outcome (i.e., daily opioid use for past 30 days). Two OARSCM participants, one of which terminated the interview before completion, and zero TAU with MyMAT participants did the 1-month follow-up interview.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | OARSCM | TAU With MyMAT
Number analyzed (Participants) | 2 | 0
Days | 0 (0) |

7. Secondary Outcome: Longest Duration of Abstinence - Phase 2 RCT (Month 3)
Description: Longest duration of consecutive days of abstinence (composite of biochemical & self-report data)
Time Frame: 3 months from participant's enrollment
Population: Participants who did not answer the follow-up call were considered lost to follow-up and assigned the worse possible outcome (i.e., daily opioid use for past 30 days). One OARSCM participant and zero TAU with MyMAT participants did the 3-month follow-up interview.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | OARSCM | TAU With MyMAT
Number analyzed (Participants) | 1 | 0
Days | 0.86 (3.93) |
Statistical Analysis 1: Comparison: OARSCM vs TAU With MyMAT; Test type: Superiority; p = 1.00, z statistics — Statistical significance was set at p<0.05. z-score = 0.329

8. Secondary Outcome: Longest Duration of Abstinence - Phase 2 RCT (Month 6)
Description: Longest duration of consecutive days of abstinence (composite of biochemical & self-report data)
Time Frame: 6 months from participant's enrollment
Population: Participants who did not answer the follow-up call were considered lost to follow-up and assigned the worse possible outcome (i.e., daily opioid use for past 30 days). Zero participants from both arms did the 6-month follow-up interview.
Arm/Group | OARSCM | TAU With MyMAT
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | OARSCM | TAU With MyMAT
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

LIMITATIONS AND CAVEATS:
Low enrollment and lack of subject response to follow-up interviews led to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT05180669/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT05180669/SAP_001.pdf